CLINICAL TRIAL: NCT00588562
Title: Rare Kidney Stone Consortium Registry for Hereditary Kidney Stone Diseases
Brief Title: Rare Kidney Stone Consortium Patient Registry
Acronym: RKSC
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Oxalosis and Hyperoxaluria Foundation (OHF) (Other)
Responsible Party: Principal Investigator, John Lieske, M.D., Mayo Clinic
Other Study IDs: 11-001702; 1U54DK083908-01 (NIH)
Record Dates: First submitted 2007-12-27; First posted 2008-01-08 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Primary Hyperoxaluria; Dent Disease; Cystinuria; APRT Deficiency
Keywords: PH; PH1; PH2; PH3; PHI; PHII; PHIII; PH NonI-NonII; Primary Hyperoxaluria; Primary Oxalosis; Hyperoxaluria; Oxalate; Cystinuria; Cystine; APRT; Adenine phosphoribosyl transferase deficiency; Dent disease; Dent
MeSH Terms: conditions — Hyperoxaluria, Primary; Dent Disease; Cystinuria; Adenine phosphoribosyltransferase deficiency; Hyperoxaluria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Primary Hyperoxaluria patients: Registry will include data on patients with confirmed diagnosis of Primary Hyperoxaluria.
- Dent Disease Patients: Registry will include data on patients with confirmed diagnosis of Dent Disease.
- Cystinuria Patients: Registry will include data on patients with confirmed diagnosis of Cystinuria.
- APRT deficiency Patients: Registry will include data on patients with confirmed diagnosis of APRT deficiency.

SUMMARY:
The purpose of this study is to collect medical information from a large number of patients in many areas of the world with primary hyperoxaluria (PH), Dent disease, Cystinuria and APRT deficiency. This information will create a registry that will help us to compare similarities and differences in patients and their symptoms. The more patients we are able to enter into the registry, the more we will be able to understand the Primary Hyperoxalurias,Dent disease, cystinuria and APRT and learn better ways of caring for patients with these diseases.

DETAILED DESCRIPTION:
This study involves the collection of medical information to create a computer database or registry for patients with PH, Dent disease, cystinuria and APRT deficiency. The information will be entered into the registry by your physician or health care provider. The computer web site for the registry is secure and protected by a required password. Some information which will be entered may include your age at first symptoms of PH,Dent disease, cystinuria or APRT, laboratory values, kidney function and the progress of your health over time. Information for an individual patient can only be viewed by the appropriate physician or staff. Once the information is entered into the registry, you will only be identified by a code number.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must have a definitive diagnosis of Primary Hyperoxaluria, Dent Disease, Cystinuria or APRT Deficiency.
* Individuals have a family history of a sibling with Primary Hyperoxaluria,Dent Disease, Cystinuria or APRT Deficiency.

Exclusion Criteria:

* Individuals who do not have Primary Hyperoxaluria, Dent Disease, Cystinuria or APRT Deficiency.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Primary Hyperoxaluria, Dent Disease, Cystinuria and APRT Deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 730 (Estimated)
Dates: Start 2003-07; Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Establish and expand registries and collaborate with patient organizations for the rapid dissemination of knowledge | Yearly
  The patient Registries will expand knowledge of the clinical expression of these disease by systematically accumulating and analyzing information regarding a larger number of patients than have been studied to date.

SECONDARY OUTCOMES:
Improved understanding of symptoms and progression of four major diseases of hereditary nephrolithiasis. | Yearly
  The goal of the patient Registries is to collect data about these rare diseases, provide a better understanding of these four conditions and help to develop new treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn S. Milliner, M.D., Principal Investigator — Primary Hyperoxaluria Registry - Mayo Clinic, Rochester, MN; David Goldfarb, MD, Study Director — Cystinuria Registry, New York University, NY; John C Lieske, MD, Study Director — Dent Disease Registry, Mayo Clinic, Rochester, MN; Vidar Edvardsson, MD, Study Director — APRT Registry, Landspitali University Hospital, Iceland
Locations (4):
- United States (3):
  - Dent Disease Registry -Mayo Clinic, Rochester, Minnesota
  - Primary Hyperoxaluria Registry - Mayo Clinic, Rochester, Minnesota
  - Cystinuria Registry - New York University, New York, New York
- APRT Registry - Landspitali Universtiy Hospital, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: Yes
Using limited data set, data will be shared through the Data Monitoring and Coordinating Center of the Rare Diseases Clinical Research Network.